CLINICAL TRIAL: NCT00325039
Title: TOMUS-Trial Of Mid-Urethral Slings
Acronym: TOMUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carelon Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK58229
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-12

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence, Stress; Surgery
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): retropubic mid-urethral sling (TVT) The specific TVT used was the Tension-free Vaginal Tape (Gynecare)
  Interventions: Procedure: retropubic mid-urethral sling (TVT)
- 2 (Active Comparator): transobturator mid-urethral sling (TVT-O and the Monarc) Two transobturator slings were used: the Tension-free Vaginal Tape Obturator (Gynecare), which is placed starting inside the vagina and coming out through the obturator foramen ("in-to-out") or the Monarc (American Medical System), which is placed starting in the groin area, passing through the obturator foramen, and then into the vagina ("out-to-in").
  Interventions: Procedure: transobturator mid-urethral sling (TVT-O and the Monarc)

INTERVENTIONS:
Procedure: retropubic mid-urethral sling (TVT) — This trial is a comparison of two types of mid-urethral slings. The retropubic mid-urethral mesh sling is used for treatment of stress incontinence; this procedure was less invasive than the fascial sling procedures that were reference standards at the start of the study. Specifically, a synthetic tape is passed transvaginally at the midurethral level through the retropubic space.
  Arms: 1
Procedure: transobturator mid-urethral sling (TVT-O and the Monarc) — This trial is a comparison of two types of mid-urethral slings. The transobturator mid-urethral sling is used for treatment of stress incontinence; this procedure was developed to minimize the potential for bladder and bowel injuries associated with the retropubic sling, since the sling is passed through the obturator canal, avoiding the pelvic organs in the retropubic space.
  Arms: 2

SUMMARY:
The primary aim of this clinical trial is to compare treatment success for two minimally invasive surgical procedures to treat stress urinary incontinence in women. These procedures are called mid-urethral slings. The secondary aims of the trial are to compare other outcomes for the two surgical procedures, including quality of life, sexual function, satisfaction with treatment outcomes, complications, and the need for other treatments(s) after surgery. Follow-up will be a minimum of two years.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Stress urinary incontinence (SUI) as evidenced by all of the following:
* Self-reported stress-type urinary incontinence symptoms, of duration ≥ 3 months
* Medical, Epidemiological and Social Aspects of Aging (MESA) stress symptom score (percent of total possible stress score) greater than MESA urge symptom score (percent of total possible urge score)
* Observation of leakage by provocative stress test at a bladder volume ≤ 300ml
* Bladder capacity ≥ 200ml by stress test
* Post-void residual (PVR) ≤ 100cc with pelvic organ prolapse (POP) Stage I or lower. If POP is Stage II-IV, PVR >100cc but ≤ 500cc is allowed
* Eligible for both retropubic and transobturator procedures
* No medical contraindications, e.g., current urinary tract infection (UTI), history of pelvic irradiation, history of lower urinary tract cancer
* American Society of Anesthesiologists (ASA) class I, II, or III
* No current intermittent catheterization
* Available for 24-months of follow-up and able to complete study assessments, per clinician judgment
* Signed consent form

Exclusion Criteria:

* Age <21 years
* Non-ambulatory (ambulatory with assistive devices does not exclude the patient)
* Pregnancy by self-report or positive pregnancy test, or self-reported intention to ever become pregnant
* Current chemotherapy or current or history of pelvic radiation therapy
* Systemic disease known to affect bladder function (i.e., Parkinson's disease, multiple sclerosis, spina bifida, spinal cord injury or trauma)
* Urethral diverticulum, current or previous (i.e. repaired)
* Prior augmentation cystoplasty or artificial sphincter
* Implanted nerve stimulators for urinary symptoms
* History of synthetic sling for stress urinary incontinence
* <12 months post-partum
* Laparoscopic or open pelvic surgery <3 months*
* Current evaluation or treatment for chronic pelvic pain (painful bladder syndrome)
* Participation in another treatment intervention trial that might influence the results of this trial
* Need for concomitant surgery requiring an abdominal incision, use of graft material in the anterior compartment, or any use of synthetic graft material
* Enrollment in other urinary incontinence trials including SISTEr/E-SISTEr or BE-DRI/E-BE-DRI

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gormley, M.D., Study Chair — Dartmouth-Hitchcock Medical Center
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Oakwood Hospital/Cancer Center, Dearborn, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Chai TC, Huang L, Kenton K, Richter HE, Baker J, Kraus S, Litman H; Urinary Incontinence Treatment Network (UITN). Association of baseline urodynamic measures of urethral function with clinical, demographic, and other urodynamic variables in women prior to undergoing midurethral sling surgery. Neurourol Urodyn. 2012 Apr;31(4):496-501. doi: 10.1002/nau.21198. Epub 2012 Feb 29. PMID 22378483
- [Background] Nygaard I, Brubaker L, Chai TC, Markland AD, Menefee SA, Sirls L, Sutkin G, Zimmern P, Arisco A, Huang L, Tennstedt S, Stoddard A. Risk factors for urinary tract infection following incontinence surgery. Int Urogynecol J. 2011 Oct;22(10):1255-65. doi: 10.1007/s00192-011-1429-9. Epub 2011 May 11. PMID 21560012
- [Background] Richter HE, Litman HJ, Lukacz ES, Sirls LT, Rickey L, Norton P, Lemack GE, Kraus S, Moalli P, Fitzgerald MP, Dandreo KJ, Huang L, Kusek JW; Urinary Incontinence Treatment Network. Demographic and clinical predictors of treatment failure one year after midurethral sling surgery. Obstet Gynecol. 2011 Apr;117(4):913-921. doi: 10.1097/AOG.0b013e31820f3892. PMID 21422865
- [Background] Chai TC, Kenton K, Xu Y, Sirls L, Zyczynski H, Wilson TS, Rahn DD, Whitcomb EL, Hsu Y, Gormley EA. Effects of concomitant surgeries during midurethral slings (MUS) on postoperative complications, voiding dysfunction, continence outcomes, and urodynamic variables. Urology. 2012 Jun;79(6):1256-61. doi: 10.1016/j.urology.2012.02.048. Epub 2012 Apr 25. PMID 22542356
- [Background] Brubaker L, Norton PA, Albo ME, Chai TC, Dandreo KJ, Lloyd KL, Lowder JL, Sirls LT, Lemack GE, Arisco AM, Xu Y, Kusek JW; Urinary Incontinence Treatment Network. Adverse events over two years after retropubic or transobturator midurethral sling surgery: findings from the Trial of Midurethral Slings (TOMUS) study. Am J Obstet Gynecol. 2011 Nov;205(5):498.e1-6. doi: 10.1016/j.ajog.2011.07.011. Epub 2011 Jul 20. PMID 21925636
- [Background] Nager CW, Sirls L, Litman HJ, Richter H, Nygaard I, Chai T, Kraus S, Zyczynski H, Kenton K, Huang L, Kusek J, Lemack G; Urinary Incontinence Treatment Network. Baseline urodynamic predictors of treatment failure 1 year after mid urethral sling surgery. J Urol. 2011 Aug;186(2):597-603. doi: 10.1016/j.juro.2011.03.105. Epub 2011 Jun 16. PMID 21683412
- [Result] Urinary Incontinence Treatment Network (UITN). The Trial of Mid-Urethral Slings (TOMUS): Design and Methodology. J Appl Res. 2008;8(1):AlboVol8No1. PMID 24772006
- [Result] Brubaker L, Rickey L, Xu Y, Markland A, Lemack G, Ghetti C, Kahn MA, Nagaraju P, Norton P, Chang TD, Stoddard A; Urinary Incontinence Treatment Network. Symptoms of combined prolapse and urinary incontinence in large surgical cohorts. Obstet Gynecol. 2010 Feb;115(2 Pt 1):310-316. doi: 10.1097/AOG.0b013e3181cb86b2. PMID 20093904
- [Result] Nager CW, Kraus SR, Kenton K, Sirls L, Chai TC, Wai C, Sutkin G, Leng W, Litman H, Huang L, Tennstedt S, Richter HE; Urinary Incontinence Treatment Network. Urodynamics, the supine empty bladder stress test, and incontinence severity. Neurourol Urodyn. 2010 Sep;29(7):1306-11. doi: 10.1002/nau.20836. PMID 20127832
- [Result] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Result] Richter HE, Kenton K, Huang L, Nygaard I, Kraus S, Whitcomb E, Chai TC, Lemack G, Sirls L, Dandreo KJ, Stoddard A. The impact of obesity on urinary incontinence symptoms, severity, urodynamic characteristics and quality of life. J Urol. 2010 Feb;183(2):622-8. doi: 10.1016/j.juro.2009.09.083. Epub 2009 Dec 16. PMID 20018326
- [Result] Sirls LT, Tennstedt S, Albo M, Chai T, Kenton K, Huang L, Stoddard AM, Arisco A, Gormley EA. Factors associated with quality of life in women undergoing surgery for stress urinary incontinence. J Urol. 2010 Dec;184(6):2411-5. doi: 10.1016/j.juro.2010.08.019. Epub 2010 Oct 16. PMID 20952014
- [Derived] Brubaker L, Litman HJ, Kim HY, Zimmern P, Dyer K, Kusek JW, Richter HE, Stoddard A; Urinary Incontinence Treatment Network. Missing data frequency and correlates in two randomized surgical trials for urinary incontinence in women. Int Urogynecol J. 2015 Aug;26(8):1155-9. doi: 10.1007/s00192-015-2661-5. Epub 2015 Mar 24. PMID 25800900
- [Derived] Wai CY, Curto TM, Zyczynski HM, Stoddard AM, Burgio KL, Brubaker L, Rickey LM, Menefee SA; Urinary Incontinence Treatment Network*. Patient satisfaction after midurethral sling surgery for stress urinary incontinence. Obstet Gynecol. 2013 May;121(5):1009-1016. doi: 10.1097/AOG.0b013e31828ca49e. PMID 23635737
- See also: Urinary Incontinence Treatment Network Public Website — http://www.uitn.net/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between April 2006 and June 2008. Patients were recruited from nine clinical sites. TOMUS (Trial Of Mid-Urethral Slings) was conducted by the Urinary Incontinence Treatment Network (UITN), a cooperative network consisting of urologists and urogynecologists at 9 clinical centers and a biostatistical coordinating center.
Pre-assignment Details: 3521 women were screened for eligibility. 1513 did not meet inclusion criteria; 1259 were eligible for inclusion in the study but were excluded (1001 declined to participate, 258 excluded for administrative reasons). 749 women provided written consent; of these 152 were excluded (63 ineligible, 66 withdrew consent, 23 administrative reasons).
Groups:
- Retropubic (RMUS): retropubic mid-urethral sling (TVT)
- Transobturator (TMUS): transobturator mid-urethral sling (TVT-O and the Monarc)
Period: Overall Study
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Started | 298 | 299
Completed | 280 | 285
Not Completed | 18 | 14
Not completed — Lost to Follow-up | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS) | Total
Number analyzed (Participants) | 298 | 299 | 597
Age, Continuous [Mean (Standard Deviation); unit: Yrs] | 52.7 (10.5) | 53.1 (11.5) | 52.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 299 | 597
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 298 | 299 | 597

OUTCOME MEASURES:

1. Primary Outcome: Objective Treatment Success at 12 Months
Description: Objective treatment success: negative stress test, negative pad test, and no retreatment for stress urinary incontinence (SUI) including behavioral, pharmacologic or surgical procedures
  A provocative stress test standardized to volume and position is performed for direct observation of urine leakage. Observed urine loss from the urethra coincidental with the Valsalva maneuver or cough is a positive test; a negative test indicates no urine loss. Pad testing quantifies the amount of urine involuntarily lost and is used to reflect everyday incontinence; it is negative if loss is <15g/24 hrs.
Time Frame: 12 months
Population: Because the study was designed as an equivalence trial, the outcome was assessed only in women treated per-protocol (n=291 and n=292 in RMUS, TMUS, respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Number analyzed (Participants) | 291 | 292
percentage of participants | 80.8 | 77.7
Statistical Analysis 1: Comparison: Retropubic (RMUS) vs Transobturator (TMUS); With 294 women/arm, the study would have 80% power to show equivalence between the two procedures, with an equivalence margin of +/- 12 percentage points, at a two-sided significance level of 5%. A planned time-to-event interim analysis of the primary outcome (objective treatment success) was conducted when 33% of the anticipated treatment failures occurred. We adjusted the primary outcome analysis for this interim look by assigning nominal alpha values of 0.049 to the 95% confidence intervals; Test type: Non-Inferiority or Equivalence — This study was an equivalence trial and was designed to have 80% power to show equivalence between the two sling procedures, with an equivalence margin of +/- 12 percentage points, at a two-sided significance level of 5%. The margin of +/- 12 was chosen on the basis of clinical considerations and a calculation of the number of patients it was feasible to enroll in the trial; difference in success rate (RMUS-TMUS) = 3.0, 95% CI 2-sided [-3.6 to 9.6]

2. Secondary Outcome: Patient Satisfaction at 12 Months
Description: Patient satisfaction was assessed at the 12 month visit with the questions, "how satisfied or dissatisfied are you with the result of bladder surgery related to urine leakage?" Possible responses were completely satisfied, mostly satisfied, neutral, mostly dissatisfied, and completely dissatisfied. Completely and mostly satisfied were reported as "satisfied" and neutral, most dissatisfied and completely dissatisfied as "not satisfied".
Time Frame: Follow-Up
Population: This is the number of women who answered the satisfaction questions at the 12 month visit (n=280 attended the 12 month visit in the retropubic arm and n=285 in the transobturator arm)
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Number analyzed (Participants) | 262 | 261
percentage of participants analyzed | 85.9 | 90.0
Statistical Analysis 1: Comparison: Retropubic (RMUS) vs Transobturator (TMUS); Although the primary aim of the study was designed as an equivalence trial, the secondary aims were considered as superiority tests; Test type: Superiority or Other; p = 0.14, Chi-squared — This was not adjusted for multiple comparisons; the a priori threshold for statistical significance was 0.05; Difference in proportions = -4.1

3. Primary Outcome: Subjective Treatment Success at 12 Months
Description: Absence of self-reported symptoms of stress-type urinary incontinence, as assessed with the use of the Medical, Epidemiological and Social Aspects of Aging (MESA) questionnaire (responded never to all 9 MESA questions), no leakage recorded in a 3-day voiding diary and no retreatment for stress incontinence including behavioral, pharmacologic or surgical treatment.
Time Frame: 12 months
Population: Because the study was designed as an equivalence trial, the outcome was assessed only in women treated per-protocol (n=291 in the Retropubic arm and n=292 in the transobturator arm).
Measure: Number; unit: percentage of participants
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Number analyzed (Participants) | 291 | 292
percentage of participants | 62.2 | 55.8
Statistical Analysis 1: Comparison: Retropubic (RMUS) vs Transobturator (TMUS); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; difference in success (RMUS - TMUS) = 6.4, 95% CI 2-sided [-1.6 to 14.3]

4. Secondary Outcome: Change in Quality of Life From Baseline to 12 Months
Description: Scores on the Incontinence Impact Questionnaire range from 0 to 400 with higher scores indicating greater impact. The scores are changes from baseline to the 12 month visit (baseline - 12 months).
Time Frame: Baseline - 12 months
Population: These are the number of patients with available quality of life data at the 12 month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Number analyzed (Participants) | 264 | 263
units on a scale | 126.8 (94.5) | 132.9 (97.8)
Statistical Analysis 1: Comparison: Retropubic (RMUS) vs Transobturator (TMUS); The null hypothesis is that the two arms do not differ according to quality of life, as measured by the IIQ; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

5. Secondary Outcome: Bother as Measured by the Urogenital Distress Inventory (UDI) at 12 Months
Description: Urogenital Distress Inventory (UDI) scores range from 0 to 300 with higher scores indicating greater distress. Scores are changes from baseline to the 12 month visit (baseline - 12 months)
Time Frame: 12 months
Population: This is the number of participants who had complete UDI information at the 12 month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Number analyzed (Participants) | 264 | 263
units on a scale | 106.7 (48.0) | 110.3 (51.2)
Statistical Analysis 1: Comparison: Retropubic (RMUS) vs Transobturator (TMUS); The UDI measure was compared using a two-sample t test; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Consistent with the primary outcome reported at 12 months, adverse event data through the 12 month visit are reported here.
Arm/Group | Retropubic (RMUS) | Transobturator (TMUS)
Serious Adverse Events (participants affected / at risk) | 41/298 | 19/299
Other Adverse Events (participants affected / at risk) | 110/298 | 89/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retropubic (RMUS) (N=298) | Transobturator (TMUS) (N=299)
Mesh exposure (Surgical and medical procedures) | 9 (10) | 5 (5)
Mesh erosion (Surgical and medical procedures) | 1 (1) | 1 (1)
Surgical site infection (Surgical and medical procedures) | 0 (0) | 2 (2)
Granulation tissue (Surgical and medical procedures) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Surgical and medical procedures) | 15 (15) | 0 (0)
Vaginal epithelial perforation (Surgical and medical procedures) | 6 (6) | 13 (13)
Recurrent cystitis, leading to diagnostic cystoscopy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolus (Vascular disorders) | 0 (0) | 1 (1)
Postoperative bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neurologic symptoms (Nervous system disorders) | 1 (1) | 0 (0)
Voiding dysfunction requiring surgery, use of catheter or both (Renal and urinary disorders) | 8 (9) | 0 (0)
Urothelial abrasion (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retropubic (RMUS) (N=298) | Transobturator (TMUS) (N=299)
Mesh exposure (Surgical and medical procedures) | 4 (4) | 3 (3)
Surgical site infection (Surgical and medical procedures) | 2 (2) | 2 (2)
Genitourinary (Renal and urinary disorders) | 40 (46) | 24 (27)
Vascular or hematologic (Vascular disorders) | 18 (20) | 7 (7)
Neurologic symptom of numbness (Nervous system disorders) | 6 (8) | 7 (9)
Neurologic symptom of weakness (Nervous system disorders) | 7 (7) | 21 (22)
Voiding dysfunction (Renal and urinary disorders) | 10 (16) | 4 (5)
Self-reported pain 6 or more weeks after procedure (General disorders) | 7 (7) | 6 (7)
New urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Persistent urge incontinence (Renal and urinary disorders) | 36 (54) | 30 (55)
Granulation tissue (Surgical and medical procedures) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Thrush (General disorders) | 1 (1) | 0 (0)
Wound edge separation (Surgical and medical procedures) | 1 (1) | 0 (0)
Minor wound (Surgical and medical procedures) | 1 (1) | 0 (0)
Medication reaction (General disorders) | 0 (0) | 1 (1)
Skin irritation (General disorders) | 0 (0) | 1 (1)
Sac in pelvis (seroma) (Renal and urinary disorders) | 0 (0) | 1 (1)
Bilateral leg pain (General disorders) | 0 (0) | 1 (1)
Decreased bladder sensation (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No